CLINICAL TRIAL: NCT04841551
Title: Kybella for the Treatment of Flank Fat (FF)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Beer, Kenneth R., M.D., PA (Individual)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KybellaFlanks 001
Record Dates: First submitted 2021-03-24; First posted 2021-04-12 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Adiposity
Keywords: kybella; flank fat
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: Single center, single arm open label treatment group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Kybella Flanks (Other): 10 subjects will be treated with Kybella in the flanks
  Interventions: Drug: Kybella Flanks

INTERVENTIONS:
Drug: Kybella Flanks — 10 subjects will be treated with Kybella in the flanks

SUMMARY:
To Determine the safety and Effectiveness of Kybella for the treatment of Flank Fat (FF)

DETAILED DESCRIPTION:
This is a single center study of the safety and efficacy of Kybella for the treatment of subcutaneous adipose in the flank area (flank fat).

Each qualified subject will undergo treatment with Kybella in the flank region for the reduction of flank fat.. Prior to treatment, the principal investigator will evaluate the severity of the subcutaneous adipose deposition of the flanks. Subjects will also have an MRI of the flanks at screening and week 12. .. Flank digital images will be taken prior to treatment and at each subsequent visit. The subjects will complete a safety and injection site response (ISR) diary beginning on the evening of treatment.

The subjects will return at Week 6 for additional treatment if warranted by the treating investigator. Subjects will be contacted via a phone call within 72 hours after each injection. Subjects will be seen at Week 6, 10, 12 and 18 (EOS) after initial treatment, at which time the subject will undergo photography and the investigator will rate treatment improvement (GAIS). The investigator will evaluate the treatment area for any adverse events (AEs). MRI study will be done at screening and at week 12.

The subject will return 6 weeks after initial treatment, and the principal investigator will determine if a touch-up treatment is warranted. If deemed necessary, a touch-up treatment may be administered Digital photography will be captured prior to treatment and following treatment. The subject will return 4 weeks after the touch-up to undergo digital photography and for the principal investigator to assess safety/improvement.

After initial treatment routine follow-up visits for safety and effectiveness will occur at Week 6, 10, 12, and 18 (EOS). A phone call will occur within 72 hours following injection. At all follow-up visits, digital photography will be captured and the investigator will rate treatment improvement (GAIS).. At screening and at Week 6, 10, 12 and 18 (EOS) subjects will complete the satisfaction of flank region questionnaire.

The goal of this study will be to assess the feasibility and efficacy of injecting Kybella for the treatment of subcutaneous fat of the flank region.

ELIGIBILITY:
Inclusion Criteria:The following are requirements for entry into the study:

1. Male or female, 21 years and above
2. Has mild to moderate flank fat
3. Written informed consent has been obtained
4. Written Authorization for Use and Release of Health and Research Study Information has been obtained
5. Written documentation has been obtained in accordance with the relevant country and local privacy requirements, where applicable.
6. Ability to follow study instructions and likely to complete all required visits
7. If the subject is a female of childbearing potential (sexually active and not sterile, surgically sterilized, or postmenopausal for at least 1 year), have a urine pregnancy test evaluated as negative within 10 days prior to enrollment, have used contraception for at least 30 days prior to enrollment, and agree to use a reliable method of contraception for the duration of the study. Pregnancies that occur during the clinical trial will be followed by the sponsor until delivery or termination.
8. Subject agrees to abstain from any treatment to the flank region including botulinum toxins, hyaluronic acid fillers, cosmetic surgery, laser/light therapy, chemical peels, etc for the duration of the study.

   -

Exclusion Criteria:

The following are criteria for exclusion from participating in the study:

1. Uncontrolled systemic disease
2. Severe cardiovascular disease
3. Known allergy or sensitivity to the study medication(s) or its components
4. Females who are pregnant, nursing, or planning a pregnancy. If a pregnancy occurs during the study the pregnancy will be followed by the sponsor until delivery or termination.
5. Current enrollment in an investigational drug or device study or participation in such a study within 30 days of entry into this study and for the duration of the study.
6. Previous treatment to the flanks with hyaluronic acid fillers or semi-permanent filler (i.e. Radiesse) in the past 12 months and for the duration of the study
7. Any use of permanent filler materials such as Artefill or silicone in the flanks.
8. Subjects planning a cosmetic procedure in the treatment area during the study period or with prior cosmetic procedures (i.e. surgery) in the treatment area or visible scars that may affect the evaluation.
9. Any subjects with volume deficit due to trauma, abnormalities in adipose tissue related to immune-mediated diseases such as generalized lipodystrophy (e.g., juvenile dermatomyositis), partial lipodystrophy (e.g., Barraquer-Simons syndrome), inherited disease, or HIV-related disease.
10. Infection or dermatoses at the injection site.
11. Evidence of recent alcohol or drug abuse.
12. Medical and/or psychiatric problems that are severe enough to interfere with the study results.
13. Known bleeding disorder or is receiving medication that will likely increase the risk of bleeding as the result of injection.
14. Has hair that would interfere with evaluation and treatment of the flank area
15. Has a tendency to develop hypertrophic scarring
16. Has a history of anaphylaxis or allergy to lidocaine (or any amide-based anesthestics), HA products, or Streptococcal protein.
17. Has porphyria
18. Has an active inflammation, infection, cancerous or precancerous lesion, or unhealed wound in the flank area.
19. Subject has a condition or is in a situation which in the Investigator's opinion may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study -

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-07-22 (Actual); Primary Completion 2022-03-02 (Actual); Study Completion 2022-03-02 (Actual)

PRIMARY OUTCOMES:
Primary effectiveness measure | Week 6, Week 10
  The change in the appearance and rating of the flank fat through MRI study and as measured by the independent observer GAIS rating. Change in the Global Aesthetic Improvement Scale (GAIS) as measured by the principal investigator. The investigator will independently assess the subject's level of improvement on the GAIS scale, comparing the live subject with his/her pre-treatment digital image, at all follow-up visits.
  5-Point Global Aestheic Improvement Scale (GAIS) Score Grade Description 2 Much Improved Marked improvement in appearance
  1 Improved Improvement in appearance, but a touch-up or re-treatment is needed 0 No Change The appearance is essentially the same as the original condition
  * 1 Worse The appearance is worse than the original condition
  * 2 Much Worse The appearance is much worse than the original condition

SECONDARY OUTCOMES:
Secondary effectiveness measure | Week 6, Week 10, Week 12
  The secondary effectiveness measure is subject responses to the subject Satisfaction with a GAIS Scoring system.
  5-Point Global Aestheic Improvement Scale (GAIS) Score Grade Description 2 Much Improved Marked improvement in appearance
  1 Improved Improvement in appearance, but a touch-up or re-treatment is needed 0 No Change The appearance is essentially the same as the original condition
  * 1 Worse The appearance is worse than the original condition
  * 2 Much Worse The appearance is much worse than the original condition

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Beer, M.D., Principal Investigator — Research Institute of the Southeast, LLC
Locations (1):
- Kenneth Beer, MD, PA, West Palm Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR
Time Frame: July 2022

REFERENCES:
- [Background] Pham CT, Lee A, Sung CT, Choi F, Juhasz M, Mesinkovska NA. Adverse Events of Injectable Deoxycholic Acid. Dermatol Surg. 2020 Jul;46(7):942-949. doi: 10.1097/DSS.0000000000002318. PMID 31977503
- [Background] Lin MJ, Dubin DP, Schwarcz RM, Khorasani H. The Impact of Submental Deoxycholic Acid Injections on Neck Surgery. J Drugs Dermatol. 2019 Dec 1;18(12):1281. PMID 31860219